CLINICAL TRIAL: NCT03817879
Title: A Randomized Controlled Study Comparing the VivaSight Double-lumen Tube With a Conventional Double-lumen Tube in Adult Patients Undergoing Thoracic Surgery
Brief Title: Double-lumen Tubes (DLT) - Health Economic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ambu A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CIS-009
Record Dates: First submitted 2019-01-09; First posted 2019-01-28 (Actual); Results first posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2019-10

CONDITIONS: Single Lung Ventilation; Thoracic Surgery; Anesthesia; Cost-effectiveness
MeSH Terms: interventions — One-Lung Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VivaSight double-lumen tube (Experimental)
  Interventions: Procedure: VivaSight double-lumen tube for single-lung ventilation
- Conventional double-lumen tube (Active Comparator)
  Interventions: Procedure: Conventional double-lument tube for single-lung ventilation

INTERVENTIONS:
Procedure: VivaSight double-lumen tube for single-lung ventilation — Procedure using a tube with a camera
  Arms: VivaSight double-lumen tube
Procedure: Conventional double-lument tube for single-lung ventilation — Procedure using a tube without a camera
  Arms: Conventional double-lumen tube

SUMMARY:
The aim of this study is to make a health economic evaluation comparing novice physicians use of VivaSight double-lumen tube and a conventional double-lumen tube for single-lung ventilation during thoracic surgery at a teaching hospital. The hypothesis is, that both double-lumen tubes are equally cost-effective and the the incidence of fiberoptic bronchoscope use it the same for both tubes.

DETAILED DESCRIPTION:
A randomized, controlled single-centre investigation comparing the VivaSight double-lumen tube and the conventional double-lumen tube at a teaching hospital. A pilot study including up to 10 subjects will be performed prior to the investigation is initiated. The investigation will include a total of 50 adult subjects (25 subjects in each group) admitted to the investigational site with established indication of single lung ventilation.

The objective of the investigation is to compare the number of times the tube position needs to be verified with a scope and relevant costs between VivaSight double lumen tube and conventional double lument tube in a cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Oral explanation of the investigation and Patient Information has been given to the subject or legal representative
* The subject or legal representative has signed the Informed Consent
* The subject is admitted at Odense University Hospital (OUH), department V
* Subjects evaluated as eligible for single-lung ventilation with the use of a left sided DLT
* Subjects > 18 years of age

Exclusion Criteria:

* Subjects with known tracheobronchial anatomic anomalies
* Subjects going for emergency procedures
* Subjects with anticipated difficult airways
* Subjects with known tracheal pathology
* Subjects requiring rapid sequence induction
* Surgeries in which other lung isolation devices or techniques may be warranted (e.g. tracheostomy, nasal intubation, bronchial blockers)
* Subjects who cannot be intubated with a double-lumen tube (VivaSight-DL or conventional DLT)
* Subjects requiring a right-sided DLT
* Subjects who had participated in the study before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will described in groups

REFERENCES:
- [Background] Larsen S, Holm JH, Sauer TN, Andersen C. A Cost-Effectiveness Analysis Comparing the VivaSight Double-Lumen Tube and a Conventional Double-Lumen Tube in Adult Patients Undergoing Thoracic Surgery Involving One-Lung Ventilation. Pharmacoecon Open. 2020 Mar;4(1):159-169. doi: 10.1007/s41669-019-0163-y. PMID 31297752

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VivaSight Double-lumen Tube | Conventional Double-lumen Tube
Started | 35 | 35
Completed | 30 | 22
Not Completed | 5 | 13
Not completed — Drop out | 5 | 12
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VivaSight Double-lumen Tube | Conventional Double-lumen Tube | Total
Number analyzed (Participants) | 30 | 22 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.80 (10.02) | 68.50 (7.16) | 66.94 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 17 | 10 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] | 172.47 (9.32) | 172.77 (9.56) | 172.60 (9.33)
Weight [Mean (Standard Deviation); unit: kg] | 74.73 (19.14) | 76.23 (17.12) | 75.37 (18.15)
Surgical lung [Count of Participants; unit: Participants]
  Left | 9 | 4 | 13
  Right | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Times Bronchoscope is Used
Time Frame: During procedure, up to 4 hours
Measure: Mean (Standard Deviation); unit: Reported uses of bronchoscopes
Arm/Group | VivaSight Double-lumen Tube | Conventional Double-lumen Tube
Number analyzed (Participants) | 30 | 22
Reported uses of bronchoscopes | 0.07 (0.25) | 3.14 (1.58)

2. Secondary Outcome: Intubation Time
Time Frame: During procedure, up to 4 hours
Reporting Status: Not Posted

3. Secondary Outcome: Number of Intubation Attempts
Time Frame: During procedure, up to 4 hours
Reporting Status: Not Posted

4. Secondary Outcome: Number of Time the Tube Was Repositioned
Time Frame: During procedure, up to 4 hours
Reporting Status: Not Posted

5. Secondary Outcome: Number of Times Repositioning of the Tube Was Prevented
Time Frame: During procedure, up to 4 hours
Reporting Status: Not Posted

6. Secondary Outcome: Cost Per Procedure
Time Frame: An average of 1 year
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Obtain User Perspective of the Device (VivaSight Double Lumen Tube or Conventional Double Lumen Tube) Used During Procedure.
Description: Qualitative assessment (face-validated and testet during pilot test) using a five-point scale (1: very easy/very good, 3: acceptable, 5: very difficult/very poor)
Time Frame: During procedure, up to 4 hours
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Patient Reported Post Operative Outcomes
Description: Qualitative assessment (face-validated and testet during pilot test) using a questionnaire registrering postoperative outcomes (Yes/No) and degree of postoperative outcomes (mild/moderate/severe)
Time Frame: Within 48 hours after the procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 48 hours post procedure.
Arm/Group | VivaSight Double-lumen Tube | Conventional Double-lumen Tube
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/22
Other Adverse Events (participants affected / at risk) | 0/30 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT03817879/Prot_SAP_000.pdf